CLINICAL TRIAL: NCT06201169
Title: Comparative Study of PEEK Bar Versus Titanium Bar Fabricated by CAD-CAM in Mandibular Hybrid Prostheses
Brief Title: PEEK Bar Versus Titanium Bar Fabricated by CAD-CAM in Mandibular Hybrid Prostheses: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amr Azab Abd El-Fattah (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Amr Azab Abd El-Fattah, assiatant lecturer, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: REC 02-21 4
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Edentulous Jaw
Keywords: Hybrid prosthesis, Polyether-ether-ketone,
MeSH Terms: conditions — Jaw, Edentulous

STUDY DESIGN:
Intervention Model Description: completely edentulous mandibular arch opposing natural dentition were selected
Who Masked: Participant, Outcomes Assessor
Masking Description: each participant enrolled in the study randomly and the results of both groups were serialized and assessed by the outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (control) (Active Comparator): The bars are fabricated from titanium. the participants received implant supported hybrid prosthesis with CAD/CAM fabricated titanium bars
  Interventions: Procedure: implant placement
- group II (Experimental): The bars are fabricated from PEEK . the participants received implant supported hybrid prosthesis with CAD/CAM fabricated PEEK bars
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — All patients received four implants in the lower arch

SUMMARY:
CAD/CAM-fabricated PEEK bar exhibited greater dimensional deviation in comparison to its titanium counterpart. Nevertheless, patients with PEEK bars reported higher satisfaction levels and lower marginal bone loss when compared to those with titanium bars.

DETAILED DESCRIPTION:
Fourteen patients with completely edentulous mandibular arch opposing natural dentition were selected and divided into two groups, seven patients in each. All patients received implant-supported hybrid prostheses with a bar fabricated by CAD/CAM milling technique. In group I (control), bar was fabricated from titanium, while in group ӀӀ, the bar was fabricated from PEEK. The evaluation of the study was done at 6 and 12 follow-up periods according to the following: 1- Experimentally by Geomagic (Geomagic, Japan) to detect any dimensional deviation of PEEK bars compared to titanium bars. 2-Clinically by questionnaire to evaluate the patient satisfaction. 3- Radiographically (digital periapical) to measure marginal bone loss around the implants.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous mandibular arch for at least six months have almost of the natural teeth in the maxillary arch with a ranged of age from 40- 60 years old.

and normal class Ӏ maxilla-mandibular relationship with a minimum 12-15 mm inter-arch space

Exclusion Criteria:

* All patient had systemic disorders that may influence soft or hard tissue healing were excluded as:

  * History of radiation therapy in the head and neck region.
  * Active infection or inflammation or flabby tissue in the mandibular arch
  * Bone diseases as osteoporosis.
  * Clenching or bruxism, temporomandibular joint troubles
  * Neurological or psychiatric handicap conditions that could interfere with good oral hygiene.
  * Heavy smoking and drug abusing

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Radiographically (digital periapical) | six and twelve months
  marginal bone loss around the implants

CONTACTS AND LOCATIONS:
Overall Officials: Research Ethics committee, Principal Investigator — Tanta University
Locations (2):
- Egypt (2):
  - Faculty of dentistry tanta university, Al Gharbī Bahjūrah, Tanta
  - Tanta University, Al Gharbī Bahjūrah, Tanta

IPD SHARING:
Plan to Share IPD: No